CLINICAL TRIAL: NCT01092117
Title: A Pivotal Clinical Study to Evaluate the Safety and Effectiveness of the Ovation™ Abdominal Stent Graft System
Brief Title: Clinical Study of the TriVascular Ovation™ Abdominal Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 771-0006
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: abdominal; aortic; aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ovation™ Abdominal Stent Graft System (Other): Implant of Ovation™ Abdominal Stent Graft System
  Interventions: Device: Ovation™ Abdominal Stent Graft System

INTERVENTIONS:
Device: Ovation™ Abdominal Stent Graft System — Implant of Ovation™ Abdominal Stent Graft System

SUMMARY:
The primary objectives of this study are to determine whether the Ovation Abdominal Stent Graft System is a safe and effective method of treating abdominal aortic aneurysms (AAA's) in those patients considered to be suitable candidates for open surgical repair.

DETAILED DESCRIPTION:
This is a Phase II prospective, consecutive enrolling, non-randomized multi-center clinical evaluation of the safety and effectiveness of the Ovation Abdominal Stent Graft System when used in the treatment of patients with AAA (Treatment Group) as compared to a performance goal (Control Group).

150 study patients will be enrolled at up to 40 institutions. An additional 100 study patients will be enrolled in the continued access phase.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Inclusion Criteria

All patients must meet all of the following inclusion criteria to be eligible for enrollment into this study:

1. Patient is > 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient is considered by the treating physician to be a candidate for elective open surgical repair of the abdominal aortic aneurysm (AAA) (i.e., category I, II, or III per American Society of Anesthesiology (ASA) classification. ASA category IV patients may be enrolled provided their life expectancy is greater than 1 year.
5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:

   * Abdominal aortic aneurysm ≥5.0 cm in diameter
   * Aneurysm has increased in size by 0.5 cm in last 6 months.
   * Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment
6. Patient has patent iliac or femoral arteries that allow endovascular access with the TriVascular Ovation Abdominal Stent Graft System.
7. Patient has a suitable non-aneurysmal proximal aortic neck length of ≥ 7 mm inferior to the most distal renal artery ostium.
8. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥10 mm. The resultant repair should preserve patency in at least one hypogastric artery.
9. Patient has a suitable non-aneurysmal proximal aortic neck luminal diameter between 16 and 30 mm.
10. Patient has suitable non-aneurysmal distal iliac luminal diameters between 8 and 20 mm.
11. Patient meets the following anatomic criteria: the distance from the most distal renal artery to most superior internal iliac artery measurement is at least 13 cm.
12. Patient has juxtarenal aortic neck angulation ≤ 60º if proximal neck is ≥10 mm and ≤ 45º if proximal neck is <10 mm.
13. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria

Patients that meet ANY of the following are not eligible for enrollment into the study:

1. Patient has a dissecting aneurysm
2. Patient has an acutely ruptured aneurysm
3. Patient has an acute vascular injury
4. Patient has a need for emergent surgery
5. Patient has a known thoracic aortic aneurysm or dissection.
6. Patient has a mycotic aneurysm or has an active systemic infection
7. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
8. Patient has had a myocardial infarction (MI) and/or stroke (CVA) within the past 6 months.
9. Patient has a major surgical or interventional procedure planned ≤30 days of the AAA repair.
10. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
11. Patient has history of bleeding disorders or refuses blood transfusions.
12. Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0 mg/dl
13. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
14. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG-based polymers, fluorinated ethylene propylene (FEP) or nitinol.
15. Patient has a body habitus that would inhibit X-ray visualization of the aorta
16. Patient has a limited life expectancy of less than 1 year
17. Patient is currently participating in another investigational device or drug clinical trial
18. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Mehta, MD, Principal Investigator — Albany Medical College
Locations (1):
- Community Care Physicians, Latham, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehta M, Valdes FE, Nolte T, Mishkel GJ, Jordan WD, Gray B, Eskandari MK, Botti C; A Pivotal Clinical Study to Evaluate the Safety and Effectiveness of the Ovation Abdominal Stent Graft System Investigators. One-year outcomes from an international study of the Ovation Abdominal Stent Graft System for endovascular aneurysm repair. J Vasc Surg. 2014 Jan;59(1):65-73.e1-3. doi: 10.1016/j.jvs.2013.06.065. Epub 2013 Aug 24. PMID 23978572

RESULTS

PARTICIPANT FLOW:
Period: Index Procedure to 1 Month
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 161
Completed | 160
Not Completed | 1
Not completed — Death | 1
Period: 1 Month
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 160
Completed | 157
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Period: 6 Months
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 157
Completed | 152
Not Completed | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3
Period: 12 Month
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 152
Completed | 138
Not Completed | 14
Not completed — Death | 11
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Period: Year 2
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 138
Completed | 128
Not Completed | 10
Not completed — Death | 5
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Period: Year 3
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 128
Completed | 109
Not Completed | 19
Not completed — Death | 7
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 3
Period: Year 4
Arm/Group | Ovation™ Abdominal Stent Graft System
Started | 109
Completed | 93
Not Completed | 16
Not completed — Death | 8
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ovation™ Abdominal Stent Graft System
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 149
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 111
  Germany | 30
  Chile | 20
American Society of Anesthesiology (ASA) Grade [Count of Participants; unit: Participants] — ASA I: A normal healthy patient without any systemic disease, undergoing elective surgery ASA II: A patient with mild systemic disease. Disease does not affect daily activities.
  ASA III: Individual with multiple system disease or well controlled major system disease. Disease does limit daily activities.
  ASA IV: Individual in imminent danger of death. Surgery is viewed to be last resort at salvaging life. Individual not expected to live through the next 24 hours.
  Participants
    ASA Grade I | 9
    ASA Grade II | 45
    ASA Grade III | 96
    ASA Grade IV | 11
Cardiovascular Disease [Count of Participants; unit: Participants]
  Coronary artery disease | 72
  Valvular heart disease | 19
  Angina | 11
  Cardiomyopathy | 11
  Congestive Heart Failure | 12
  Myocardial infarction | 33
  Arrhythmia | 35
  Hypertension | 136
  Hypotension | 1
  Hyperlipidemia | 113
Peripheral Vascular Disease, Stroke and Aneurysm History [Count of Participants; unit: Participants]
  Peripheral vascular disease | 38
  Carotid artery disease | 21
  Transient ischemic attack | 8
  Stroke (CVA) | 13
  Family History of aneurysms | 10
Pulmonary History [Count of Participants; unit: Participants]
  Smoking | 113
  Chronic obstructive pulmonary disease (COPD) | 44
Gastrointestinal, Genitourinary, Reproductive History [Count of Participants; unit: Participants]
  Renal failure/insufficiency | 22
  Diabetes | 34
  Alcohol abuse | 3
Hematological Problems (hemorrhage, coagulopathy disorder, anemia, platelet disorder) [Count of Participants; unit: Participants] | 12
Other Significant Medical Condition [Count of Participants; unit: Participants] | 122
Proximal Aorta [Mean (Standard Deviation); unit: mm] — Proximal Neck Length Defined by orthogonal CT cross section immediately distal to the lowest lying renal artery measuring ≥3 mm and, by definition, continues until the aortic diameter changes by >10%.
  mm
    Aortic diameter 35 mm proximal to proximal renal artery | 25.0 (2.7)
    Aortic diameter at distal renal artery | 22.5 (2.7)
    Aortic diameter 7 mm distal to distal renal artery | 22.1 (2.9)
    Aortic diameter 13 mm distal to distal renal artery | 22.7 (3.1)
    Proximal neck length | 23.0 (12.5)
Proximal Aorta-Juxtarenal angle [Mean (Standard Deviation); unit: Degrees] | 19.1 (13.5)
Aortic Aneurysm-Aortic aneurysm diameter [Mean (Standard Deviation); unit: mm] — Proximal Neck Calcification and Thrombus Scoring Amount of calcium and / or thrombus present in the cross-sectional area of the target location of the sealing ring (IR+4 to IR+10).
  mm | 53.6 (9.0)
Aortic aneurysm diameter distribution [Count of Participants; unit: Participants]
  40.0mm-49.9mm | 57
  50.0mm-59.9mm | 81
  60.0mm-69.9mm | 14
  70.0mm-79.9mm | 5
  80.0mm-89.9mm | 2
  90.0mm-99.9mm | 2
Distal Aorta [Mean (Standard Deviation); unit: mm]
  Aortic bifurcation diameter | 20.3 (6.9)
  Left iliac diameter | 13.7 (3.3)
  Left iliac minimum access diameter | 7.0 (1.6)
  Right iliac diameter | 13.9 (3.0)
  Right iliac minimum access diameter | 7.0 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint is Defined as the Percentage of Subjects Who Experience a Major Adverse Event Within 30 Days of the Initial Procedure.
Description: Major adverse events (MAE) are defined as any one of the following events:
  * Death
  * Myocardial Infarction
  * Stroke (excludes TIA)
  * Renal Failure (excludes renal insufficiency)
  * Respiratory Failure (excludes COPD or pulmonary complications)
  * Paralysis (excludes paraparesis)
  * Bowel Ischemia
  * Procedural Blood Loss (≥1,000 cc)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation™ Abdominal Stent Graft System
Number analyzed (Participants) | 161
Participants | 4

2. Primary Outcome: The Primary Effectiveness Endpoint is Percentage of Subjects That Achieve Treatment Success.
Description: Treatment Success is a composite endpoint assessed at 12 months that requires the following criteria to be met:
  * Technical Success, defined as successful delivery and deployment of one aortic body and two iliac limbs.
  * Freedom from Type I & III endoleaks at 12 months
  * Freedom from stent graft migration at 12 months
  * Freedom from abdominal aortic aneurysm (AAA) enlargement at 12 months
  * Freedom from abdominal aortic aneurysm (AAA) rupture and conversion to open repair through 12 months
  Endoleak Definition:
  Type I - Ineffective seal at either the proximal or distal sealing zones Type II - Retrograde blood flow from lumbar arteries, the inferior mesenteric artery, or other collateral vessels into the aneurysm sac Type III - A leak caused by fabric tears or disruption, component disconnection, or graft disintegration Type IV - Blood flow through an intact fabric.
Time Frame: 1 year
Population: 138 subjects completed study through 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation™ Abdominal Stent Graft System
Number analyzed (Participants) | 138
Participants | 137

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Ovation™ Abdominal Stent Graft System
All-Cause Mortality (participants affected / at risk) | 35/161
Serious Adverse Events (participants affected / at risk) | 129/161
Other Adverse Events (participants affected / at risk) | 144/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ovation™ Abdominal Stent Graft System (N=161)
Hematoma (Blood and lymphatic system disorders) | 4
Post-procedureal Bleeding (Blood and lymphatic system disorders) | 4
Acute Blood Loss (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Disseminated Intravascular Coagulation with Septic Shock (Blood and lymphatic system disorders) | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1
Elevated White Blood Cells (Blood and lymphatic system disorders) | 1
Heparin Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1
Lymphatic leak (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Polycythaemia Vera (Blood and lymphatic system disorders) | 1
Severe Anemia Secondary To Myelodisplasia (Blood and lymphatic system disorders) | 1
Subararchnoidal Bleeding (Blood and lymphatic system disorders) | 1
Angina (Cardiac disorders) | 6
Arrhythmia (Cardiac disorders) | 7
Congestive Heart Failure (Cardiac disorders) | 10
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 3
Myocardial Infarction (Cardiac disorders) | 6
Atrial fibrillation with RVR (Cardiac disorders) | 1
Atrial fibrillation With Rapid Ventricular Response (Cardiac disorders) | 1
Aortic Valve Stenosis (Cardiac disorders) | 3
Cardiac Arrest (Cardiac disorders) | 2
Cardiogenic Shock (Cardiac disorders) | 1
Coronary Artery Disease: Chest Pain, Le Edema, Ruq Abdominal Pain (Cardiac disorders) | 1
Mitral Reguritation (Cardiac disorders) | 1
Severe Aortic Stenosis (Cardiac disorders) | 1
Sinoatrial Node Dysfunction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tricuspid Regurgitation (Cardiac disorders) | 1
Unstable Angina (Cardiac disorders) | 1
Worsening Atrial Fibrillation (Cardiac disorders) | 2
Worsening Chronic Heart Disease (Cardiac disorders) | 1
Worsening Congestive Heart Failure (Cardiac disorders) | 1
Thyreoidectomy (Endocrine disorders) | 1
Circulatory Disorder Left Eye (Eye disorders) | 1
Surgical Procedure: pars-Plana Vitrectomy, Cerclage and Kryocoagulation right Eye (Eye disorders) | 1
Adynamic ileus (Gastrointestinal disorders) | 1
Bowel ischemia (Gastrointestinal disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Infection (other than wound) (Gastrointestinal disorders) | 8
Acute On Chronic Pancreatitis (Gastrointestinal disorders) | 1
Air in Intestine (Gastrointestinal disorders) | 1
Bleeding Duodenal Ulcer (Gastrointestinal disorders) | 1
Bloody Stools (Gastrointestinal disorders) | 1
Bowel Perforation (Gastrointestinal disorders) | 1
Cholecystitis (Gastrointestinal disorders) | 2
Choledocholithiasis (Gastrointestinal disorders) | 1
Cholelithiasis (Gastrointestinal disorders) | 1
Dilated Biliary Ducts (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Duodenal Angiodysplasia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastrointenstinal Bleed (Gastrointestinal disorders) | 5
Hematochezia (Gastrointestinal disorders) | 1
Hemorrhoids With Hematochezia (Gastrointestinal disorders) | 1
Ischemic Colitis (Gastrointestinal disorders) | 1
Nausea W/ Vomiting (Gastrointestinal disorders) | 1
Urinary Retention (Gastrointestinal disorders) | 3
Fever (Gastrointestinal disorders) | 2
Bilateral Leg Weakness (General disorders) | 1
Chest Pain (General disorders) | 1
Chest Tightness/Non-Cardiac Chest Pain (General disorders) | 2
Collapse (General disorders) | 1
Death (General disorders) | 1
Death from unknown cause (General disorders) | 2
Dizziness (General disorders) | 1
Epigastric/Substernal Pain (General disorders) | 1
Groin Pain (General disorders) | 1
Groin Pain Inguinal Hernia (General disorders) | 1
Leg Pain (General disorders) | 1
Lightheaded (General disorders) | 1
Lower Extremity Edema (General disorders) | 1
Lumbar And Right Lower Extremity Severe Pain (General disorders) | 1
Near Syncope/Weakness (General disorders) | 1
Necrosis (General disorders) | 1
Right Lower Extremity Significant Swelling W/Edema (General disorders) | 1
Right Upper Quadrant Pain (General disorders) | 1
Syncope (General disorders) | 3
Abdominal and Chest Pain (General disorders) | 1
Syncope Related To Blood Loss From Chest Wall Hematoma (General disorders) | 1
Unknown at this time- awaiting hospital records (General disorders) | 1
Worsening Claudication (General disorders) | 1
Worsening Lower Back And Leg Pain (General disorders) | 1
Anaphylactic Shock (Immune system disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Abdominal Sepsis (Infections and infestations) | 1
Acute Pyelonephritis (Infections and infestations) | 1
C-Diff Infection (Infections and infestations) | 1
Erysipel (Infections and infestations) | 1
Fungal Infection In Groin (Infections and infestations) | 1
Herpes Zoster, Left Lumbar Pain And Echymosis (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Pneumonia-MRSA (Infections and infestations) | 1
Respiratory Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic Right Knee Joint (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Spontaneous Bacterial Peritonitis (Infections and infestations) | 1
Urinary Tract Infection By Hydronephrosis (Infections and infestations) | 1
Viral Encephalopathy (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Lactic Acidosis With Liver Failure (Metabolism and nutrition disorders) | 1
Severe Hyponatremia (Metabolism and nutrition disorders) | 1
Broken Shoulder (Musculoskeletal and connective tissue disorders) | 1
Effusion of the left hip (Musculoskeletal and connective tissue disorders) | 1
Fall-fx R prox humerous (Musculoskeletal and connective tissue disorders) | 1
Fracture right hip (Musculoskeletal and connective tissue disorders) | 2
Hip fracture (Musculoskeletal and connective tissue disorders) | 1
J1 DJD L hip (Musculoskeletal and connective tissue disorders) | 1
L1 Compression Fracture (Musculoskeletal and connective tissue disorders) | 1
Left hip fracture (Musculoskeletal and connective tissue disorders) | 1
Left knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1
R Knee Arthroplasty (Musculoskeletal and connective tissue disorders) | 1
R Knee spacer removal (Musculoskeletal and connective tissue disorders) | 1
Right femur fracture (Musculoskeletal and connective tissue disorders) | 1
Acute Gout Left Knee (Musculoskeletal and connective tissue disorders) | 1
Acute Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1
Acute Onset Of Chronic Polyarthitis (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Elective Right Total Hip Arthroplasty (Musculoskeletal and connective tissue disorders) | 1
Gait Weakness/Progressive Decline (Musculoskeletal and connective tissue disorders) | 1
Groin Hernia (Metabolism and nutrition disorders) | 1
Hernia (Musculoskeletal and connective tissue disorders) | 1
Incarcerated L Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 2
Incarcerated Left Inguinal Hernia With Secondary small bowel obstruction (Musculoskeletal and connective tissue disorders) | 1
Rupture Tendons Right Shoulder. Arthroscopic Repair (Musculoskeletal and connective tissue disorders) | 1
artificial Knee joint (Musculoskeletal and connective tissue disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 2
endoprothesis of right knee (Musculoskeletal and connective tissue disorders) | 1
enstage cuff tear arthrop (Musculoskeletal and connective tissue disorders) | 1
fractured left hip (Musculoskeletal and connective tissue disorders) | 1
hip-tep surgery right (Musculoskeletal and connective tissue disorders) | 1
hip/back pain (Musculoskeletal and connective tissue disorders) | 1
impingement-syndrome (Musculoskeletal and connective tissue disorders) | 1
lumbal spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis, right hip (Musculoskeletal and connective tissue disorders) | 1
Pain left knee (Musculoskeletal and connective tissue disorders) | 1
Quadricept tendon rupture (Musculoskeletal and connective tissue disorders) | 1
Right knee revision (Musculoskeletal and connective tissue disorders) | 1
Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Bladder Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mass In Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastic Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Nasal Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peritoneal Carcinosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Brenner Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Prostatic Hypertrophy With Obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperechoic Mass Lesions Noted Throughout The Liver with hepatomegaly (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
L Thyroid Mass With Thyroid Lobectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Poylp-Hyperplastic And 3 Tubular Adenomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Colon Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Recurrent Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Recurrent Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vallecular Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urotheluim Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vesical Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular Accident/Stroke (Nervous system disorders) | 5
Acute Encephalopathy (Nervous system disorders) | 1
Concussion, Laceration (Nervous system disorders) | 1
Encepalopathy, Multifactorial (Nervous system disorders) | 1
New Onset Idiopathic Seizures (Nervous system disorders) | 1
Subacute Subdural Hematoma (Nervous system disorders) | 1
Worsening Seizures (Nervous system disorders) | 1
Transient Ischemic Attack (TIA) (Nervous system disorders) | 3
Device Fracture (Product Issues) | 3
Illac Limb Occlusion (Product Issues) | 5
Indeterminate (Product Issues) | 1
Polymer Leak (Product Issues) | 1
Type IA (Proximal) (Product Issues) | 4
Type IB (Distal) (Product Issues) | 1
Type II (Product Issues) | 6
Wound Infection (Product Issues) | 1
Acute Psychosis (Psychiatric disorders) | 1
Acute Severe Anxiety (Psychiatric disorders) | 1
Acute Severe Depression (Psychiatric disorders) | 1
Altered Mental Status (Psychiatric disorders) | 1
Anxiety/Restlessness (Psychiatric disorders) | 1
Change In Mental Status - Cerebral Cramps And Coma (Psychiatric disorders) | 1
Dementia (w/ Hospitalization) (Psychiatric disorders) | 1
Hospital Admission to Rearrange Psychiatric Medications (Psychiatric disorders) | 1
Worsening Mental Status (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 3
Anuria (Renal and urinary disorders) | 1
Dj Stent Change (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Kidney Stone (Renal and urinary disorders) | 1
Kidney Stones/Rt Flank Pain/Er Visit (Renal and urinary disorders) | 1
Pre-Existing Renal Insufficiency Hospitalization (Renal and urinary disorders) | 2
Renal Stone (w/ Admission) (Renal and urinary disorders) | 1
Ureteral Surgery (Renal and urinary disorders) | 1
Left Orchyepididimitis, Right Epididimitis (Reproductive system and breast disorders) | 1
Right Testis Hydrocele Surgical Repair (Reproductive system and breast disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 11
Acute Hypercapnic And Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5
Acute Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Chest Stab Wound (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (COPD) Exacerbation (Respiratory, thoracic and mediastinal disorders) | 8
End Stage Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxiemia/Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Episode of Heavy Dispnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion, Kard. Decompensation (Respiratory, thoracic and mediastinal disorders) | 1
Progression Of Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure Secondary to COPD (Respiratory, thoracic and mediastinal disorders) | 1
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis With Dizziness And Flashing Lights (Respiratory, thoracic and mediastinal disorders) | 1
Spontaneous Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Weakness And Increase Oxygen Demand (Respiratory, thoracic and mediastinal disorders) | 1
Worsening COPD And Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Worsening Respiratory Failure Secondary To Septic Shock and MRSA Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Chest Wall Hematoma (Skin and subcutaneous tissue disorders) | 1
Cutaneous Rash (Skin and subcutaneous tissue disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Endographic Repair Of Known Thoracic Penetrating Ulcer (Skin and subcutaneous tissue disorders) | 1
Hematoma Left Arm (Skin and subcutaneous tissue disorders) | 1
Hematoma Left Thigh, Wound Healing Disorder (Skin and subcutaneous tissue disorders) | 1
Left Lower Extremity Cellulitis (Skin and subcutaneous tissue disorders) | 1
Necrosis Of Right Toe (Skin and subcutaneous tissue disorders) | 1
Open Wound, Necrosis (Skin and subcutaneous tissue disorders) | 1
Right Hip Incision And Drainage (Skin and subcutaneous tissue disorders) | 2
Stage 3 Pressure Ulcer Bilateral Buttocks (Skin and subcutaneous tissue disorders) | 1
Ulcera Cruris With Known Paod Iv (Skin and subcutaneous tissue disorders) | 1
Attempted Suicide (Social circumstances) | 1
Mechanical Fall (Social circumstances) | 1
Numerous Falls resulting in Hospitalization (Social circumstances) | 1
Small Subarachnoid Hemorrhage Due To Fall (Social circumstances) | 1
Allergic To Contrast Agent (Surgical and medical procedures) | 1
Elective Prostatectomy (Surgical and medical procedures) | 1
Medication Induced Encephalopathy, Diagnosed With orthostatic hypotension (Surgical and medical procedures) | 1
Post-surgical Hematoma, Hydrocele Repair (Surgical and medical procedures) | 1
Post-Procedural Hematuria (Surgical and medical procedures) | 1
Postoperative Compartment Syndrome Of Rt. Leg Due to Hematoma (Surgical and medical procedures) | 1
Aneurysm enlargement (Vascular disorders) | 4
Aneurysm rupture (Vascular disorders) | 1
Aortic Body Stenosis (Vascular disorders) | 1
Peripheral Ischemia (Vascular disorders) | 3
Ae Code L13. Other Vascular- Supra-Renal Vs. Celiac Aneurysm Rupture (Vascular disorders) | 1
Aneurysm Enlargement Due To Type Ii Endoleak (Vascular disorders) | 1
Aneurysm Expand Without Endoleak (Vascular disorders) | 1
Aneurysm Spurium Of Left Arm (Vascular disorders) | 1
Ascending Aortic Aneurysm (Vascular disorders) | 1
Bilateral Pulmonary Emboli (Vascular disorders) | 1
Claudication (L) Lower Extremity; (L) Stenosis & Urinary retention (Vascular disorders) | 1
Extrinsic Compression Aortic Body (Vascular disorders) | 1
N2 Left Carotid Endarterectomy (Vascular disorders) | 1
N2 Right Carotid Endarterectomy (Vascular disorders) | 1
Pseudoaneurysm (Vascular disorders) | 1
Pulmonary Hypertension (Vascular disorders) | 1
Rt Sfa Occlusion (Vascular disorders) | 1
Superior Mesenteric Vein Occlusion (Vascular disorders) | 1
Supra Renal Aneurysm Rupture (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 1
Venous Insufficiency (Vascular disorders) | 1
Worsening Perivascular Disease (Vascular disorders) | 1
Vascular Occlusion (Vascular disorders) | 3
Vascular Trauma (Vascular disorders) | 2
Renal Failure (Renal and urinary disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ovation™ Abdominal Stent Graft System (N=161)
Coagulopathy (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Anemia Due To B12 Deficiency (Blood and lymphatic system disorders) | 1
Anemia-Low Hemoglobin And Hematocrit (Blood and lymphatic system disorders) | 1
Anemia-Macrocytic (Blood and lymphatic system disorders) | 1
Decreased Hematocrit Level (Blood and lymphatic system disorders) | 1
Elevated Inr Levels (Blood and lymphatic system disorders) | 1
Elevated Wbc (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 3
N2- Worsening Of Anemia Post Op (Blood and lymphatic system disorders) | 1
Supratherapeutic Inr 8.6 (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina (Cardiac disorders) | 7
Arrhythmia (Cardiac disorders) | 4
Congestive Heart Failure (Cardiac disorders) | 5
Acute Congestive Heart Failure (Cardiac disorders) | 1
Afib With Rapid Ventricular Response (Cardiac disorders) | 1
Apical Thrombus (Cardiac disorders) | 1
Asymptomatic Pvc's During Routine Colonoscopy (Cardiac disorders) | 1
Atrial Septal Aneurysm (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Decreased Ef From 35% To 25% (Cardiac disorders) | 1
High Pulse Rate- Tachycardia (Cardiac disorders) | 1
Increase Troponin Levels (Cardiac disorders) | 1
Irregular Heart Beat (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Pfo (Congenital, familial and genetic disorders) | 1
Hearing Loss (Ear and labyrinth disorders) | 1
Hearing Loss Left Ear (Ear and labyrinth disorders) | 1
Otitis Media/Hearing Loss (Ear and labyrinth disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 1
Diabetes (Endocrine disorders) | 1
Diabetic Ketacedosis (Endocrine disorders) | 1
Elevated Tsh (Endocrine disorders) | 1
Exacerbation Of Type Ii Diabetes (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Increased Glucose Level (Endocrine disorders) | 1
Positive Ketones In Urine (Endocrine disorders) | 1
Blurred Vision R Eye (Eye disorders) | 1
Ambulatory Elective Cataract Op (Eye disorders) | 1
Bruised Left Eye (Eye disorders) | 1
Cataract In Left Eye (Eye disorders) | 2
Cataract Phacoemulsification Of The Left Eye. (Eye disorders) | 1
Cataract Phacoemulsification Of The Right Eye (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctivitis Right Eye (Eye disorders) | 1
Incisional Biopsy Of Left Upper Eyelid (Eye disorders) | 1
Macular Degeneration (Eye disorders) | 1
Occular Rosacea (Eye disorders) | 1
Removal Of Cataracts (Eye disorders) | 1
Cataract Right Eye (Eye disorders) | 3
Adynamic ileus (Gastrointestinal disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
"stomach Gnawing" (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Barrett's Esophagus (Gastrointestinal disorders) | 1
Barrett's High Grade Dysplasia (Gastrointestinal disorders) | 1
Blood In Stool (Gastrointestinal disorders) | 1
Bloody Stools (Gastrointestinal disorders) | 1
Cholitis With Urinary Retention And Rectal Urgen (Gastrointestinal disorders) | 1
Colon Polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 1
Diverticulosis (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Esophageal Spasm (Gastrointestinal disorders) | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
Gi Bleeding With Esophagil Varicosis (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Irregular Bowel Movements (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Nausea And Vomiting. Etiology (Gastrointestinal disorders) | 2
Pancreatic Head Lesion (Gastrointestinal disorders) | 1
Sigma Diverticulosis (Gastrointestinal disorders) | 2
Upper Gi Bleed (Gastrointestinal disorders) | 1
Upper Gi Endoscopy - Multiple Thermal Ablation O (Gastrointestinal disorders) | 1
Fever (General disorders) | 4
1+ Edema Bilat Lower Extremities (General disorders) | 1
1+ Pitting Edema (General disorders) | 1
Abdominal Pain (General disorders) | 1
Allergic Reaction To Klonopin (General disorders) | 1
Arm Pain (General disorders) | 1
Atypical Chest Pain. All Cardiac Diagnostic -Neg (General disorders) | 1
Back Pain (General disorders) | 5
Bilateral Leg Fatigue (General disorders) | 1
Bilateral Lower Extremity Edema (General disorders) | 3
Bilateral Lower Leg Pain (General disorders) | 1
Bruising Of Right Upper Arm (General disorders) | 1
Burning Feeling In Chest (General disorders) | 1
C/O Hip Pain (General disorders) | 1
Calf Pain (General disorders) | 1
Chest And Back Pain (General disorders) | 1
Chest Pain (General disorders) | 1
Chest Pressure (General disorders) | 1
Deconditioning (General disorders) | 1
Difficulty Sleeping (General disorders) | 1
Dizziness (General disorders) | 3
Epistaxis (General disorders) | 2
Fall At Home (General disorders) | 3
False Aneurysma Right Inguinal Side (General disorders) | 1
Fatigue (General disorders) | 2
Groin Pain (General disorders) | 2
Heache/Nausea (General disorders) | 2
Increasingly Swollen Lower Extremities (General disorders) | 1
Intermittent Groin Pain (General disorders) | 3
Intractable Hiccups (General disorders) | 1
Laceration Left Thumb (General disorders) | 1
Left Flank Pain (General disorders) | 1
Left Leg Swelling (General disorders) | 1
Left Lower Extremity Edema (General disorders) | 1
Left Lower Leg And Ankle 2+ Pitting Edema (General disorders) | 1
Legs Feel "rubbery" (General disorders) | 1
Lower Back And Leg Pain (General disorders) | 1
Malaise- General (General disorders) | 1
N2: Pain In Both Inguinal (General disorders) | 1
Nausea (General disorders) | 1
Night Sweats (General disorders) | 1
Pain In Kidney Area (General disorders) | 1
Pain In The Right Upper Quadrant Of Abdomen (General disorders) | 1
Patient Went To Er For Abdominal Pain (General disorders) | 1
Poor Sleep (General disorders) | 1
Progressive Lower Limb Weakness (General disorders) | 1
Psa-Values Increased (General disorders) | 1
Right Ear Pain (General disorders) | 1
Right Flank Pain (General disorders) | 1
Right Groin Pain (General disorders) | 1
Right Hip Pain (General disorders) | 2
Right Side Stitch (General disorders) | 1
Right Upper Quadrant Abdominal Pain (General disorders) | 1
Rt Groin Site Swollen And Burning With Hard Lump (General disorders) | 1
Sob While Walking (General disorders) | 1
Soreness In Chest (General disorders) | 1
Syncope (General disorders) | 2
Weakness (General disorders) | 1
Worsening Of Lower Extremity Edema (General disorders) | 1
Worsening of Restless Leg Syndrome (General disorders) | 1
Wound Discomfort (General disorders) | 1
Infection (other than wound) (Infections and infestations) | 14
Cellulitis Left Lower Extremity (Infections and infestations) | 1
Helicobacter Pylori (Infections and infestations) | 1
Mrsa Bacteremia (Infections and infestations) | 1
N2- Herpes Zoster With Postherpetic Neuralgia (Infections and infestations) | 1
Recurrent Left Lower Extremity Cellulitis (Infections and infestations) | 1
Right Lower Extremity Infection (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Sinus Infection (Infections and infestations) | 1
Subclinical Shingles Outbreak (Infections and infestations) | 1
Tooth Absess (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Urinary Tract Infection Due To Chronic Indwelling Foley Catheter (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 3
Calcium Level Remains Below Normal At 8.2 (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Low Vitamin D (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Paraproteinemia Protein 10.2 (Metabolism and nutrition disorders) | 1
Protein Malnutrition (Metabolism and nutrition disorders) | 1
Unintentional Weight Loss (Metabolism and nutrition disorders) | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Carpal Tunnel Injection (Musculoskeletal and connective tissue disorders) | 1
Carpal Tunnel sundrome (Musculoskeletal and connective tissue disorders) | 1
DDD lower spine (Musculoskeletal and connective tissue disorders) | 1
Foot drop (Musculoskeletal and connective tissue disorders) | 1
Lt. knee pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain Shoulder (Musculoskeletal and connective tissue disorders) | 1
Rt knee pain, torn tissue (Musculoskeletal and connective tissue disorders) | 1
Rt achilles injury/tear (Musculoskeletal and connective tissue disorders) | 1
Rt hip pain (Musculoskeletal and connective tissue disorders) | 1
Rt knee pain- arthritis (Musculoskeletal and connective tissue disorders) | 1
Acute Synovitis (Musculoskeletal and connective tissue disorders) | 1
Advanced Tooth Carie With Acute Pain (Musculoskeletal and connective tissue disorders) | 1
Bilateral Hernia Inguinal Hernia Repair (Musculoskeletal and connective tissue disorders) | 1
Bilateral Inguinal Hernias (Musculoskeletal and connective tissue disorders) | 1
Bursitis Olecrani Right Side (Musculoskeletal and connective tissue disorders) | 1
Compression Injury Upper Thoracic Spine Vertebra (Musculoskeletal and connective tissue disorders) | 1
Dental Caries With Lip Ulcer (Musculoskeletal and connective tissue disorders) | 1
Exacerbation Of Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 1
Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 1
Left Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 1
Lumbar Spondylosis, Lumbar Facet Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal- Myalgias (Musculoskeletal and connective tissue disorders) | 1
Pain Upper Leg And Sural Muscle (Musculoskeletal and connective tissue disorders) | 1
Right Inguinal Hernia Incarceration (Musculoskeletal and connective tissue disorders) | 1
Right Knee/Calf Numbness (Musculoskeletal and connective tissue disorders) | 1
Sprained Left Wrist/Inflammatory Arthritis (Musculoskeletal and connective tissue disorders) | 1
T12 compression fracture (Musculoskeletal and connective tissue disorders) | 1
Thoracic Vertebra broken (Musculoskeletal and connective tissue disorders) | 1
Torn right rotator cuff (Musculoskeletal and connective tissue disorders) | 1
compression fx vertebrae (Musculoskeletal and connective tissue disorders) | 1
left achilles tendinosis (Musculoskeletal and connective tissue disorders) | 1
left hip pain (Musculoskeletal and connective tissue disorders) | 1
leg pain (Musculoskeletal and connective tissue disorders) | 1
osteoarthritis Rt knee (General disorders) | 1
right elbow strain (Musculoskeletal and connective tissue disorders) | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Large Seroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ct Guide Lung Biopsy Of Pulmonary Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Excision Basaliom At Left Upper Arm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Generalized Intermittent Pain Secondary To Metas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Increasing Psa With Known Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paresthesia (Nervous system disorders) | 3
Benign Essential Tremor (Nervous system disorders) | 1
Bilateral Numbness In Feet (Nervous system disorders) | 1
Contusion Cerebra (Nervous system disorders) | 1
Exacerbation Of Sciatica (Nervous system disorders) | 1
Leg Weakness And Vertigo (Nervous system disorders) | 1
Mild Dementia/Memory Dysfunction/Cerebral De-Gen (Nervous system disorders) | 1
Neurologic/Musculoskeletal Pain Left Upper Extre (Nervous system disorders) | 1
Neurological Changes (Nervous system disorders) | 1
Normal Pressure Hydrocephalus (Nervous system disorders) | 1
Questionable Seizure (Nervous system disorders) | 1
Self Limited Tremor Of Head & Left Upper Limb, 1 (Nervous system disorders) | 1
Syncope, Confusion, Light Headedness (Nervous system disorders) | 1
Vertigo/Headache (Nervous system disorders) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
Device Fracture (Product Issues) | 4
Indeterminate (Product Issues) | 1
Type II Endoleak (Product Issues) | 83
Type IA (Proximal) (Product Issues) | 2
Type IIIA (Disconnectino/Disjunction) (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Dementia (Psychiatric disorders) | 3
Increasing Memory Loss (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Mild Confusion (Psychiatric disorders) | 1
Worsening Anxiety (Psychiatric disorders) | 1
Worsening Depression (Psychiatric disorders) | 1
Renal Failure (Renal and urinary disorders) | 3
Renal Insufficiency (Renal and urinary disorders) | 6
Acute Kidney Injury With High Potassium (Renal and urinary disorders) | 1
Bladder Dome Mucosal Nodule (Renal and urinary disorders) | 1
Bph (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Hydronephrosis (Renal and urinary disorders) | 1
Hypercalcemia (Renal and urinary disorders) | 1
Increased Bun Level (Renal and urinary disorders) | 2
Increased Creatinine Level (Renal and urinary disorders) | 1
Intermittent Urinary Tract Infection (Renal and urinary disorders) | 1
Kidney Infection (Renal and urinary disorders) | 2
Microhematuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Renal Masses Increase In Size (Renal and urinary disorders) | 1
Rt Kidney Cyst With Mild Thickening (Renal and urinary disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 3
Worsening Renal Insufficiency (Renal and urinary disorders) | 1
Worsening Renal Insufficiency Ckd Stage III (Renal and urinary disorders) | 1
Worsening Renal Insufficiency Ckd Stage IV (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 4
Impotence (Reproductive system and breast disorders) | 1
Right Spermocele (Reproductive system and breast disorders) | 1
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Acute Sinusitis, Maxillary (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Bibasilar Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bilateral Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4
Centrilobular And Paraseptal Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Copd (Respiratory, thoracic and mediastinal disorders) | 3
Copd Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Emphysematous Changes In Lungs (Respiratory, thoracic and mediastinal disorders) | 2
Exacerbated Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Focal Bronciolitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia And Copd Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Left Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
New 5 Mm Nodule Right Lower Lobe, Nonspecific (Respiratory, thoracic and mediastinal disorders) | 1
Non-Cardiac Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Non-Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough With Yellow Sputum (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Fibrosis- Amiodarone Related (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Nodules (Respiratory, thoracic and mediastinal disorders) | 1
Right Pleual Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Short Of Breath (Respiratory, thoracic and mediastinal disorders) | 3
Small Right Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
sob (Respiratory, thoracic and mediastinal disorders) | 1
Upper Lobe Infiltrate (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
Anterior Ankle Ulcer (Skin and subcutaneous tissue disorders) | 1
Bilat Feet Non-Healing Sores (Skin and subcutaneous tissue disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema Over Doral Aspect Of Left Foot (Skin and subcutaneous tissue disorders) | 1
Fall With Facial Abrasions (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Laceration Of Small Right Toe (Skin and subcutaneous tissue disorders) | 1
Left Foot Ulcer (Skin and subcutaneous tissue disorders) | 1
Lipoma Excision (Skin and subcutaneous tissue disorders) | 1
Mild Wound Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Petechial Rash On Shins Related To Chemotherapy (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Sebaceous Cyst Right Posterior Neck (Skin and subcutaneous tissue disorders) | 1
Skin Biopsies (Skin and subcutaneous tissue disorders) | 1
Skin Integrity (Skin and subcutaneous tissue disorders) | 1
Suspect Birthmark (Skin and subcutaneous tissue disorders) | 1
Intraoperative Bleeding (Surgical and medical procedures) | 8
Lymphocele/Lymphatic Fistula (Surgical and medical procedures) | 1
Acute Blood Loss Anemia Following Orif (Surgical and medical procedures) | 1
Bilateral Groin Erythema (Surgical and medical procedures) | 1
Cr 1.7. Ct Was Done W/O Contrast and Ultrasound (Surgical and medical procedures) | 1
Erythema Around Groin Incision (Surgical and medical procedures) | 1
Incisional Hernia After Nephrectomia (Surgical and medical procedures) | 1
Iv Dye Reaction (Surgical and medical procedures) | 1
Pain Over Acid (Surgical and medical procedures) | 1
Post Operative Anemia (Surgical and medical procedures) | 1
Post-Operative Incisional Pain (Surgical and medical procedures) | 1
Prolonged Intubation Because Of Anesthesia (Surgical and medical procedures) | 1
Reaction During Ct Scan (Surgical and medical procedures) | 1
Right Groin 1mm Opening (Surgical and medical procedures) | 1
Vancomycin Toxicity (Surgical and medical procedures) | 1
Slight Reaction To Contrast Medium (Surgical and medical procedures) | 1
Aneurysm enlargement (Vascular disorders) | 6
Aortic Body Stenosis (Vascular disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Dissection (Vascular disorders) | 2
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 10
Peripheral Ischemia (Vascular disorders) | 1
Aneurysm Enlargement (Vascular disorders) | 1
Celiac Artery Stenosis (Vascular disorders) | 2
Dissection Of Right External Iliac Artery (Vascular disorders) | 1
Dvt (Vascular disorders) | 1
Left Carotid Artery Stenosis (Vascular disorders) | 1
Left Iliac Limb Stenosis (Vascular disorders) | 1
Left Renal Artery Calcified Plaque (Vascular disorders) | 1
Left Renal Artery Stenosis (Vascular disorders) | 2
Malfunctioning Valves In Right Great Saphenous V (Vascular disorders) | 1
Multiple Peripheral Cns Emboli (Vascular disorders) | 1
Obstruction Of Illiac Arteries Without Symptoms (Vascular disorders) | 1
Petechial Hemorrhage (Vascular disorders) | 1
Progression Of Pvd Stenosis Left External Iliac (Vascular disorders) | 1
Right Carotid Stenosis (Vascular disorders) | 1
Right Common Femoral Artery Aneurysm (Vascular disorders) | 1
Right Renal Artery Stenosis (Vascular disorders) | 1
S/P Taa Endorepair Now With Type Ii Endoleak (Vascular disorders) | 1
Small Ascending Thoracic Aneurysm (Vascular disorders) | 1
Stenosis Right Renal Artery (Vascular disorders) | 1
Superficial Acute Thrombophlebitis (Vascular disorders) | 1
Superficial Phlebitis L Upper Extremity (Vascular disorders) | 1
Thoracic Aortic Aneurysm (Vascular disorders) | 2
Uncontrolled Hypertension (Vascular disorders) | 1
Worsening Claudication (Vascular disorders) | 1
Worsening Hypertension (Vascular disorders) | 1
Vascular Occlusion (Vascular disorders) | 1
Left Upper Lip Laceration (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or itsagents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. PI can publish institution's data/results 18 months after study conclusion at all sites or when multi-center results are published or notification that results will not be published. Institution is to submit drafts of manuscripts to Endologix 30 days prior to submission for publication or presentation.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-07-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT01092117/Prot_SAP_ICF_000.pdf